CLINICAL TRIAL: NCT07244692
Title: Investigation Of The Effects Of Occupational Therapy Interventions Added To Reformer Pilates Exercises In Office Workers
Brief Title: Occupational Therapy Interventions Added To Reformer Pilates Exercises In Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Raziye Şavkın, Assoc. Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-380663
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Occupational Therapy; Office Workers; Pilates Exercise
Keywords: Occupational therapy; Office workers; Reformer Pilates; Quality of life; Occupational performance
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reformer Pilates Only Group (Active Comparator): Participants in the Reformer Pilates Only Group will receive a standard reformer Pilates exercise program under the supervision of a physiotherapist for four weeks. The program will consist of eight sessions, performed twice a week.
  Each session will last 50 minutes and will include the following components:
  5 minutes of standard reformer Pilates warm-up exercises, 40 minutes of reformer Pilates exercises, 5 minutes of cool-down exercises. The exercise intensity will be progressively increased throughout the program as follows: Week 1: 8-10 repetitions, Week 2: 10-12 repetitions, Weeks 3 and 4: 12-15 repetitions.
  Interventions: Other: Reformer Pilates
- Occupational Therapy + Reformer Pilates Group (Experimental): Participants in this group will complete the same standard reformer Pilates exercise program as the comparison group. In addition, they will receive an individualized occupational therapy-based intervention program.
  The occupational therapy-based intervention program will be planned individually for each participant at the beginning of the study, based on occupations identified through the Canadian Activity Performance Scale. This program will include interventions designed to support the achievement of personalized goals in occupational performance areas such as improving ergonomic conditions in the office environment, activities of daily living, instrumental activities of daily living, leisure activities, and social participation.
  Interventions: Other: Reformer Pilates; Other: Occupational Therapy

INTERVENTIONS:
Other: Reformer Pilates — Participants in the Reformer Pilates Only Group will receive a standard reformer Pilates exercise program under the supervision of a physiotherapist for four weeks. The program will consist of eight sessions, performed twice a week.
  Each session will last 50 minutes and will include the following components: 5 minutes of standard reformer Pilates warm-up exercises, 40 minutes of reformer Pilates exercises, 5 minutes of cool-down exercises.
  The exercise intensity will be progressively increased throughout the program as follows: Week 1: 8-10 repetitions, Week 2: 10-12 repetitions, Weeks 3 and 4: 12-15 repetitions.
Other: Occupational Therapy — Participants will receive an individualized occupational therapy-based intervention program.The occupational therapy-based intervention program will be planned individually for each participant at the beginning of the study, based on occupations identified through the Canadian Activity Performance Scale. This program will include interventions designed to support the achievement of personalized goals in occupational performance areas such as improving ergonomic conditions in the office environment, activities of daily living, instrumental activities of daily living, leisure activities, and social participation.
  Arms: Occupational Therapy + Reformer Pilates Group

SUMMARY:
As computer use continues to increase, work-related musculoskeletal disorders have become a major health concern among individuals working in office environments. A lack of awareness regarding the risks of working in ergonomically unsuitable conditions contributes to the development of musculoskeletal problems due to prolonged incorrect posture. Ergonomically inadequate work environments have been reported to negatively affect employee well-being, increase musculoskeletal symptoms, and reduce work performance by affecting motivation, concentration, and other individual factors. Studies indicate that productivity losses in such conditions may range from 2.4 percent to 14.8 percent. To prevent musculoskeletal problems, reduce pain, and improve quality of life in office workers, it is recommended that the ergonomic quality of the work environment be improved and that employees be encouraged to participate in exercise programs.

The purpose of this study is to examine the effects of occupational therapy interventions added to reformer Pilates exercises in office workers. Occupational therapy interventions include ergonomic training, strategies to increase physical activity levels, and meaningful activities planned specifically for each participant. To date, to the best of our knowledge, no studies have examined the effectiveness of combining occupational therapy interventions with reformer Pilates exercises in individuals working in office settings.

It is anticipated that the integration of person-centered occupational therapy interventions with reformer Pilates exercises will lead to improvements in fatigue, burnout, and musculoskeletal symptoms, as well as enhanced quality of life in participants. In addition, occupational therapy interventions may reduce absenteeism resulting from musculoskeletal problems. Consequently, it is expected that healthcare costs may decrease while workplace productivity and efficiency may increase.

DETAILED DESCRIPTION:
Offices are environments where repetitive movements such as writing and prolonged screen use are common, often leading to poor posture, high levels of inactivity, and intensive engagement in administrative tasks. Since the mid-1980s, with the beginning of the information age, the use of computers in the workplace has increased substantially. Desktop computers, laptops, and tablets have become essential tools for communication and project management.

For office workers who spend a significant portion of their day working at a computer, the excessive load placed on the musculoskeletal system has become an important occupational ergonomics issue, contributing to the development of various musculoskeletal disorders. Risk factors related to repetitive tasks, continuous work, and poor posture are widely recognized as ergonomic risk factors.

Increasing evidence indicates that working in an ergonomically inadequate office environment can lead to musculoskeletal problems, negatively affect employee well-being, and reduce work productivity. Inadequate environmental conditions in office settings are often described as environmental stressors. Elements that determine the quality of the office environment include temperature, humidity, noise, vibration, colors, lighting, and air quality.

It has been suggested that improving factors that determine office environment quality may reduce the number of days employees take off work due to discomfort, enhance productivity, decrease stress by improving motivation, and ultimately support cost savings for organizations.

Ergonomic risk assessment approaches highlight that improper posture in office workers may result from shortcomings in workspace design or improper use of body mechanics by employees. Knowledge and awareness of ergonomics are considered protective in preventing musculoskeletal problems. Ergonomic interventions combined with principles from occupational health and safety, organizational psychology, and sociology may help better understand occupational behaviors and support workplace well-being.

In addition to ergonomic conditions, individual factors such as gender, age, education level, lifestyle habits, smoking, duration of employment, obesity, lack of exercise, and poor physical fitness also contribute to musculoskeletal disorders.

To prevent musculoskeletal problems, reduce pain, and improve quality of life in the increasing number of office workers, it is recommended to optimize workplace ergonomics and encourage employees to participate in exercise programs. Exercise-based physiotherapy approaches in office workers have been shown to reduce musculoskeletal pain symptoms and improve quality of life. Office workers who regularly engage in exercise programs generally report better overall well-being compared to those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 50,
* Having worked full-time at a desk job for at least 6 months,
* Being classified as sedentary according to the short form of the International Physical Activity Questionnaire,
* Not having previously participated in occupational therapy intervention,
* Ability to understand, speak, and write Turkish,
* Ability to understand verbal and written information provided,
* Volunteer status.

Exclusion Criteria:

* Working in a role outside the scope of office work (e.g., kitchen, cleaning, etc.),
* Having undergone surgery related to the musculoskeletal system within the last 6 months,
* The presence of any clinical or orthopedic condition that may limit the performance of Reformer Pilates exercises (malignancies, infections, inflammatory diseases, severe osteoporosis, metabolic bone diseases, pregnancy, cognitive impairment, nerve root compression, history of spinal surgery, etc.).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Cornell Musculoskeletal Discomfort Questionnaires | 10 minutes
  The Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) is used to assess the frequency, and work interference of musculoskeletal discomfort across different body regions. It helps ergonomists and health professionals identify problem areas and evaluate the impact of work tasks or interventions on employee comfort and performance.
Maslach Burnout Inventory | 10 minutes
  The Maslach Burnout Inventory is used to assess occupational burnout. The Maslach Burnout Inventory consists of three subscales and 23 items: emotional exhaustion (9 items), depersonalization (5 items), and low personal ccomplishment (8 items). The emotional exhaustion and depersonalization subscales are scored on a 5-point Likert-type scale, ranging from 0 never to 4 always, while the low personal accomplishment subscale is scored the opposite way. Possible scores for each subscale range from 0-36 for emotional exhaustion, 0-20 for depersonalization, and 0-32 for low personal accomplishment.
The Multidimensional Assessment of Fatigue | 5 minutes
  The Multidimensional Assessment of Fatigue (MAF) Scale is a self-report questionnaire designed to measure fatigue as a multidimensional experience rather than just tiredness. The scale has 16 items that measure five dimensions of fatigue: degree (item 1), severity (item 2), distress (item 3), degree of interference with activities of daily living (items 4-14), and timing (items 15-16). Items 1-14 contain 10-point numerical rating scales and items 15-16 have multiple-choice responses. The 10-point numerical rating scale ranges from 1 (not at all) to 10 (a great deal).
The World Health Organization Quality of Life Scale-BREF (WHOQOL-BREF) | 5 minutes
  The WHOQOL-BREF is a 26-item instrument consisting of four domains:physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. The physical health domain includes items on mobility, daily activities, functional capacity, energy, pain, and sleep. The psychological domain measures include self-image, negative thoughts, positive attitudes, self-esteem, mentality, learning ability, memory concentration, religion, and the mental status. The social relationships domain contains questions on personal relationships, social support, and sex life. The environmental health domain covers issues related to financial resources, safety, health and social services, living physical environment, and transportation.
AI Posture Evaluation and Correction System (APECS): Body Posture Evaluation | 5 minutes
  Digital posture evaluation with APECS uses software created for the evaluation of posture with non-invasive photogrammetry techniques and correction of postural asymmetry and disorders with various exercises. APECS is available for download in the Google Play Store. APECS performs posture assessment with markers placed on the patient's body photograph and uses algorithms to assess correct body symmetry. APECS provides a rapid analysis of anthropometric characteristics of posture. It uses standardized landmarks and anatomical angles for postural assessment. Latin names of anthropometric landmarks and a list of relevant angles are available in the application.
30-Second Sit-to-Stand Test | 30 seconds
  This test evaluates individuals' sit-to-stand activity, lower extremity strength and dynamic balance. For the test, a chair with a seat height of approximately 43,18 cm and a backrest is used, along with a stopwatch. The chair is secured to prevent movement during the sit-to-stand activity, and care is taken to ensure that the participant's feet are in contact with the floor when seated. The test involve the participant sitting comfortably on the chair with full contact for 30 seconds, then transitioning to a standing position, and finally returning to a seated position on the chair. The stopwatch is started at the moment of the first rise, and the number of sit-to-stand repetitions perform by the individual within 30 seconds is recorded.
Functional Reach Test | 5 minutes
  The functional reach test is a commonly used test for assessing dynamic balance. During the assessment, participants are asked to turn sideways to the wall, flex their arm to 90 degrees, and make a fist with their hand. In this position, the level of the third metacarpophalangeal joint is marked as the starting position, and participants are asked to reach forward as far as possible without taking a step. At the furthest point reached, the third metacarpophalangeal joint is marked again. The distance between the two marked points is recorded in centimeters. The measurement is repeated three times, and the average of the three measurements is taken.
Half Squat Test | 5-7 minutes
  The half squat test is used to assess participants' lower extremity muscular endurance. Participants are asked to assume a half-squat position on a hard surface, with their feet shoulder-width apart, arms crossed over their chest, and torso upright, without shoes. The stopwatch is started with the "Go" command, and the squatting times are recorded.
Canadian Occupational Performance Measure: COPM | 1-2 hours
  The COPM is a client-centred outcome measure for individuals to identify and prioritize everyday issues that restrict their participation in everyday living. This measure focuses on occupational performance in all areas of life, including self-care, leisure and productivity. The COPM is a semi-structured interview that enables an open dialogue between client and therapist on issues of importance to the client. COPM steps:
  1. Therapist introduction and explanation of COPM
  2. Client identifies specific activities and prioritize activities that are perceived as challenging for them
  2.Rates the current level of performance and satisfaction on a scale of 1-10 for each activity 4.Therapist and client collaborate to set client-centered goals based on identified activities 5.Therapist Documentation and intervention planning 6. Therapist Re-assessment and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Raziye Şavkın, Assoc. Prof., Study Chair — Pamukkale University; Gülden Önal, PT, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)